CLINICAL TRIAL: NCT04573504
Title: Antibiotics for Severe Perineal Laceration to Prevent Infection Following Repair
Acronym: ASPIRe
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Oluwateniola Brown, Assistant Professor, Northwestern University, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00212963
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Vaginal Laceration During Delivery
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic Group (Experimental): The antibiotic regimen chosen is based on the Royal College of Obstetricians and Gynecologists' recommendations (Augmentin and Flagyl or Clindamycin and Flagyl if they are allergic to Penicillin). The dosage for the antibiotics are the following: Flagyl 500mg po BID (twice a day) X 5 days, Clindamycin 400 mg po TID (three times a day) X 5 days, Augmentin 875mg po BID X 5 days.
  Interventions: Drug: Augmentin/Flagyl or Augmentin/Clindamycin
- Placebo Group (Placebo Comparator): Women randomized not to receive antibiotics will be given placebo tablets postpartum, so they will all have an identical experience to the women in the experimental (antibiotic) group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Augmentin/Flagyl or Augmentin/Clindamycin — Women who suffer a severe vaginal laceration at Prentice Women's Hospital will be randomized to receive 5-days of oral antibiotics or placebo pills after getting a standard one-time dose of IV antibiotics at the time of repair.
  Arms: Antibiotic Group
Drug: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
Many women experience severe anal sphincter lacerations during childbirth, which put them at risk for infection, improper healing, and accidental bowel leakage. This study aims to determine if oral antibiotics following vaginal delivery in women with severe tears can prevent wound infection and breakdown, and ultimately, accidental bowel leakage. Women who suffer a severe vaginal laceration will be randomized to receive 5-days of oral antibiotics or placebo pills after getting a standard one-time dose of IV antibiotics at the time of repair. All women will have immediate, intensive follow-up with an Urogynecologist at our well-established PEAPOD peripartum clinic at 1 week, 2 weeks, and 3 months postpartum to monitor wound healing and infection. At these visits, we also will assess women's perception of their well-being, perineal pain, and bowel symptoms. All participants will be invited to remain in the study for long-term follow-up. Our goal is to establish whether a five-day course of oral antibiotics should be a standard part of clinical care for severe postpartum lacerations.

DETAILED DESCRIPTION:
Approximately 3,000,000 women have vaginal deliveries each year in the United States.

Five percent, (i.e., 150,000) of these women will experience an obstetrical anal sphincter injury (OASIS). OASIS is associated with chronic pain and sexual dysfunction. Moreover, 25% of women with OASIS will suffer from chronic accidental bowel leakage. In other words, one new woman every 14 minutes experiences an injury that leads to uncontrollable leakage of stool and gas. This woman is not only a new mother, but she may also be a teacher, a construction worker, a nurse, a doctor, or an executive who will have to deal with this devastating and embarrassing condition for the rest of her life. At age 45, women suffer from accidental bowel leakage at a rate that is eight times higher than that of men of the same age (1).

It is likely that accidental bowel leakage is related not only to the structural disruptions that occur with OASIS, but also from complications, such as infection and poor wound healing. Women who suffer OASIS are at high risk for infection and poor healing; this is not surprising given that these lacerations are repaired and then continue to heal in a contaminated field (near stool). Poor healing and infection in the setting of OASIS make accidental bowel leakage, chronic pain, and sexual dysfunction even more likely (2-6). Unfortunately, even those infections that are recognized early and treated can still cause accidental bowel leakage decades after childbirth (7-9).

Despite the many women affected by OASIS and its debilitating ramifications through the arc of a woman's life, there is a lack of evidence-based best practice to guide treatment and follow-up when it does occur. Even though infection and poor healing compromise outcomes, there are limited data regarding best practice to prevent of these complications. The use of antibiotics at the time of OASIS repair has become common based on our division's previous studies (15-18). However, no studies have been done to determine whether oral antibiotics immediately postpartum can further decrease the incidence of short and long-term complications. The Royal College of Obstetricians and Gynecologists recommends the use of antibiotics after OASIS repair (10), however, the basis of this recommendation is founded only on expert opinion. On the other hand, the American College of Obstetricians and Gynecologists provides no recommendation with regard to whether antibiotics should be used in the postpartum time. At our institution, almost all women who sustain OASIS during vaginal delivery receive a single dose of IV antibiotics based on our previously published work at Prentice, however, that while many physicians chose to administer oral antibiotics based on expert opinions, it is unknown whether these provide any specific benefit - again as many physicians chose to administer antibiotics regardless of the evidence to date. Standard care postpartum both nationally and internationally is highly varied and likely based on physician training and preference (11).

Therefore, there is a great need for a trial to determine whether the use of supplemental antibiotics for 5 days postpartum will decrease rates of perineal wound infection and breakdown and improve maternal health outcomes. Such a trial will guide best practice, enhance the care of women, and potentially reduce the debilitating consequences of OASIS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* 3rd or 4th degree laceration upon delivering vaginally at Prentice Women's Hospital
* English-speaking
* Administered Ancef during wound repair
* First Delivery
* Single child being born
* Term Delivery (i.e. at least 37 weeks gestation)

Exclusion Criteria:

* Under 18 years old
* Non-English speaking
* Delivery of more than one fetus (i.e. twins or other multiples)
* Patient is taking systemic steroids
* Allergy to Amoxicillin AND Clindamycin
* Infant with severe jaundice who is receiving breastmilk
* Women who have medical contraindications to the use of metronidazole, clindamycin, and amoxicillin clavulanate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-09-23 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
This study has one endpoint which will be the 3-month postpartum visit and where all study participants will have completed their study questionnaires. | 2 years
  The primary outcome measure will be at the 3 month postpartum visit where all study participants have complete all study procedures and surveys. We anticipate it will take two years for all participants to have met the time frame of completing their 3 month post-partum visit.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwateniola Brown, M.D, Principal Investigator — Northwestern Medicine
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No